CLINICAL TRIAL: NCT00943852
Title: A Double-Blind, Randomized, Placebo-Controlled, 5-Period Crossover Study to Evaluate the Effects of a Single Dose of Losartan, a Single Dose of Isosorbide Mononitrate (ISMN), and Single Doses of Losartan + ISMN on Central Blood Pressure Measurements in Mildly Hypertensive Patients
Brief Title: The Effect of Losartan and Losartan Plus Isosorbide Mononitrate on Central Blood Pressure Measurements (0954-317)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0954-317; MK0954-317; 2009_610
Record Dates: First submitted 2009-07-21; First posted 2009-07-22 (Estimated); Results first posted 2010-07-15 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Losartan; isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- 1 (Active Comparator): losartan 100 mg
  Interventions: Drug: losartan potassium
- 2 (Active Comparator): ISMN 60 mg
  Interventions: Drug: Comparator: isosorbide mononitrate (ISMN)
- 3 (Active Comparator): losartan 100 mg + ISMN 15 mg
  Interventions: Drug: Comparator: losartan + ISMN
- 4 (Active Comparator): losartan 100 mg + ISMN 60 mg
  Interventions: Drug: Comparator: losartan + ISMN
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: losartan potassium — Single dose losartan 100 mg in one of five treatment periods
  Other Names: COZAAR
  Arms: 1
Drug: Comparator: isosorbide mononitrate (ISMN) — Single dose ISMN 60 mg in one of five treatment periods
  Other Names: IMDUR
  Arms: 2
Drug: Comparator: losartan + ISMN — Single dose losartan 100 mg and ISMN 15 mg in one of five treatment periods
  Arms: 3
Drug: Comparator: losartan + ISMN — Single dose losartan 100 mg and ISMN 60 mg in one of five treatment periods
  Arms: 4
Drug: Comparator: Placebo — Single dose placebo only in one of five treatment periods
  Arms: 5

SUMMARY:
This study will qualify a functional model that can measure central blood pressure and vascular compliance effects through noninvasive means.

ELIGIBILITY:
Inclusion Criteria:

* Patient is in good health with the exception of mild to moderate hypertension
* Patient is willing to comply with the study restrictions
* Patient does not smoke

Exclusion Criteria:

* Patient has a history of any illness that might confound the results of the study or make participation in the study unsafe
* Patient is taking a prescription medication that is contraindicated for use with COZAAR® or IMDUR®
* Patient has a condition for which there is a warning, contraindication, or precaution against the use of COZAAR® or IMDUR®

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-08; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Kaufman R, Nunes I, Bolognese JA, Miller DL, Salotti D, McCarthy JM, Smith WB, Herman GA, Feig PU. Single-dose effects of isosorbide mononitrate alone or in combination with losartan on central blood pressure. J Am Soc Hypertens. 2010 Nov-Dec;4(6):311-8. doi: 10.1016/j.jash.2010.10.004. PMID 21130977

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Entered: 31-Aug-2006
  Last Patient Last Visit: 11-Dec-2006
  Number of Sites: 1
Groups:
- Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN: Placebo / Losartan 100 mg / Losartan 100 mg + Isosorbide Mononitrate (ISMN) 15 mg / Losartan 100 mg + ISMN 60 mg / ISMN 60 mg - single dose with ≥ 4 days washout between doses
- Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN: Losartan 100 mg / ISMN 60 mg / Losartan 100 mg + ISMN 60 mg / Placebo / Losartan 100 mg + ISMN 15 mg - single dose with ≥ 4 days washout between doses
- ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN: ISMN 60 mg / Losartan 100 mg + ISMN 15 mg / Placebo / Losartan 100 mg / Losartan 100 mg + ISMN 60 mg - single dose with ≥ 4 days washout between doses
- Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo: Losartan 100 mg + ISMN 15 mg / Losartan 100 mg + ISMN 60 mg / Losartan 100 mg / ISMN 60 mg / Placebo - single dose with ≥ 4 days washout between doses
- Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan: Losartan 100 mg + ISMN 60 mg / Placebo / ISMN 60 mg / Losartan 100 mg + ISMN 15 mg / Losartan 100 mg - single dose with ≥ 4 days washout between doses
- Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN: Placebo / ISMN 60 mg / Losartan 100 mg / Losartan 100 mg + ISMN 60 mg / Losartan 100 mg + ISMN 15 mg - single dose with ≥ 4 days washout between doses
- Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN: Losartan 100 mg / Losartan 100 mg + ISMN 15 mg / ISMN 60 mg / Placebo / Losartan 100 mg + ISMN 60 mg - single dose with ≥ 4 days washout between doses
- ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo: ISMN 60 mg / Losartan 100 mg + ISMN 60 mg / Losartan 100 mg + ISMN 15 mg / Losartan 100 mg / Placebo - single dose with ≥ 4 days washout between doses
- Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan: Losartan 100 mg + ISMN 15 mg / Placebo / Losartan 100 mg + ISMN 60 mg / ISMN 60 mg / Losartan 100 mg - single dose with ≥ 4 days washout between doses
- Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN: Losartan 100 mg + ISMN 60 mg / Losartan 100 mg / Placebo / Losartan 100 mg + ISMN 15 mg / ISMN 60 mg - single dose with ≥ 4 days washout between doses
Period: First Period of Treatment Intervention
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period After Period 1 Treatment
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 2 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — BP too low for dosing at the next period | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Period of Treatment Intervention
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period After Period 2 Treatment
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Trial stopped early | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Third Period of Treatment Intervention
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period After Period 3 Treatment
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Did not meet criteria for next period | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Fourth Period of Treatment Intervention
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period After Period 4 Treatment
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 2 | 1 | 1 | 1 | 1 | 0 | 1 | 1 | 1 | 1
Completed | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not Completed | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Not taking medication per protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Trial stopped early | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Period: Fifth Period of Treatment Intervention
Arm/Group | Placebo / Losartan / Losartan + ISMN / Losartan + ISMN / ISMN | Losartan / ISMN / Losartan + ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Placebo / Losartan / Losartan + ISMN | Losartan + ISMN / Losartan + ISMN / Losartan / ISMN / Placebo | Losartan + ISMN / Placebo / ISMN / Losartan + ISMN / Losartan | Placebo / ISMN / Losartan / Losartan + ISMN / Losartan + ISMN | Losartan / Losartan + ISMN / ISMN / Placebo / Losartan + ISMN | ISMN / Losartan + ISMN / Losartan + ISMN / Losartan / Placebo | Losartan + ISMN / Placebo / Losartan + ISMN / ISMN / Losartan | Losartan + ISMN / Losartan / Placebo / Losartan + ISMN / ISMN
Started | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Completed | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants in Study
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 57.2 [46 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Exclusionary Medication Washout [Number; unit: participants]
  Yes | 3
  No | 10
Diastolic Blood Pressure [Mean (Full Range); unit: mm Hg] | 90.6 [77 to 103]
Heart Rate [Mean (Full Range); unit: Beats per Minute] | 75.4 [48 to 99]
Systolic Blood Pressure [Mean (Full Range); unit: mm Hg] | 141.5 [114 to 165]

OUTCOME MEASURES:

1. Primary Outcome: Mean Augmentation Index Percent Change From Baseline After Single Doses of Losartan 100 mg Plus ISMN 60 mg Versus Single Dose of Losartan 100 mg
Description: The augmentation index (AIx) is defined as the ratio of augmentation (Δ P) to central pulse pressure and expressed as percent. AIx = (ΔP/PP) x 100, where P = pressure and PP = Pulse Pressure. A mathematical transfer function translated the peripheral wave form into a central waveform using an FDA approved process based on directly recorded arterial pressure values. The mean AIx for each subject was estimated as a time-weighted average over the 10-hour post dose observation period and expressed as a change from baseline.
Time Frame: Baseline and 10 hours postdose
Population: All subjects who received single doses of losartan 100 mg + ISMN 60 mg and/or single dose of losartan 100 mg
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | Losartan 100 mg + ISMN 60 mg | Losartan 100 mg
Number analyzed (Participants) | 8 | 10
Percent Change | -24.9 (3.8) | -1.8 (3.8)
Statistical Analysis 1: Comparison: Losartan 100 mg + ISMN 60 mg vs Losartan 100 mg; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha = 0.05; Fixed effects model with terms for subject, treatment and period

2. Primary Outcome: Mean Augmentation Index Percent Change From Baseline After Single Doses of Losartan 100 mg + ISMN 60 mg Versus Single Dose of Placebo
Description: as for outcome 1
Time Frame: Baseline and 10 hours postdose
Population: All subjects who received single doses of Losartan 100 mg + ISMN 60 mg and/or single dose of placebo
Measure: Least Squares Mean (Standard Deviation); unit: Percent Change
Arm/Group | Losartan 100 mg + ISMN 60 mg | Placebo
Number analyzed (Participants) | 8 | 8
Percent Change | -24.9 (3.8) | -1.3 (3.8)
Statistical Analysis 1: Comparison: Losartan 100 mg + ISMN 60 mg vs Placebo; Test type: Superiority or Other; p < 0.001, ANOVA — 1-sided, alpha = 0.05; Fixed effects model with terms for subject, treatment and period

ADVERSE EVENTS:
Time Frame: Run-in period through 14 days post last dose of study drug (documented by telephone contact or in person)
Description: One (1) of the 13 enrolled subjects completed one period of the study and (1) of the 13 enrolled subjects completed 2 periods of the study prior to termination of the study.
  These subjects were included in the AE summary tables having been exposed to treatment, but were not included in the statistical analysis.
Arm/Group | Placebo | Losartan 100 mg | Losartan 100 mg + ISMN 15 mg | Losartan 100 mg + ISMN 60 mg | ISMN 60 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11 | 0/13 | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 2/11 | 1/13 | 4/11 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=12) | Losartan 100 mg (N=11) | Losartan 100 mg + ISMN 15 mg (N=13) | Losartan 100 mg + ISMN 60 mg (N=11) | ISMN 60 mg (N=12)
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 1
Oedema Peripheral (General disorders) | 0 | 0 | 1 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 3
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 3 | 0

LIMITATIONS AND CAVEATS:
Due to lower than expected Blood Pressure's in individual patients, an interim analysis was undertaken after 11 patients had completed 3 to 5 of the study periods; enough data was already collected to meet objectives, so the trial was stopped early.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.